CLINICAL TRIAL: NCT00669565
Title: A Phase II Safety and Efficacy Study of Bavituximab Plus Paclitaxel and Carboplatin in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Safety and Efficacy Study of Bavituximab Plus Paclitaxel and Carboplatin to Treat Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: A.J. Leyco, RN/Associate Director, Clinical Affairs, Peregrine Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0702
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Carcinoma Breast Stage IV
Keywords: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bavituximab — Receive weekly bavituximab at a dose of 3 mg/kg until disease progression, and carboplatin at a dose of AUC = 2 and paclitaxel 100 mg/m2 on days 1, 8, and 15 of a 28-day cycle for up to 6 cycles.

SUMMARY:
This is a phase II, multicenter, single-arm, open-label safety and efficacy study of bavituximab in combination with carboplatin plus paclitaxel in patients with locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Living in India for the duration of the study
* Adult females over age 18 years of age with a life expectancy of at least 3 months
* Confirmed breast cancer with evidence of locally advanced or metastatic disease
* Disease that is measurable by radiology imaging
* Ambulatory and capable of all selfcare but unable to carry out any work activities.
* Adequate laboratory results (hematologic, renal, hepatic)
* Negative pregnancy test

Exclusion Criteria:

* History of or susceptibility to bleeding or coagulopathy (e.g., von Willebrand Disease or Hemophilia)
* Any history of thromboembolic events (clots within blood vessels)
* Ongoing treatment with high doses of anticoagulants
* Use of hormone therapy
* Advanced peripheral neuropathy (e.g., numbness, tingling, and/or pain in distal extremities)
* Prior chemotherapy, immunotherapy or radiotherapy to an area of measurable disease unless disease had recurred after radiotherapy
* Radiotherapy within 2 weeks entering the study
* Chemotherapy, immunotherapy or radiotherapy within 4 weeks of starting the study
* Allergies to Polysorbate 80 or drugs containing polyoxyethylated castor oil (e.g. cyclosporine)
* Diagnosed and active CNS disease or metastatic lesions
* Major surgery within 4 weeks of starting the study
* Pregnant or nursing
* Uncontrolled disease (e.g., diabetes, hypertension, thyroid disease)
* History of heart disease
* History of any condition requiring treatment with anti-inflammatory, anti-platelet drugs or steroids
* Diagnosed with HIV or hepatitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the overall response rate (CR+PR) | Until disease progression

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - Rajalakshmi Multispecialty Hospital, Bangalore
  - Bangalore Institute of Oncology, Banglore
  - Apollo Specialty Hospitals, Chennai
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - Regional Cancer Center, Kerala
  - Medical College Hospital, Kolkata
  - Bharath Hospital and Institite of Oncology, Mysore
  - Curie Manavata Cancer Center, Nashik
  - Ruby Hall Clinic, Pune